CLINICAL TRIAL: NCT00396422
Title: A Phase IIa Randomized, Double-blind, Placebo-Controlled, Parallel Group, Multi-Center, Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of RWJ-445380 Administered to Patients With Plaque Psoriasis
Brief Title: Study to Investigate the Safety, Tolerability, Absorption, Distribution, Metabolism, and Elimination of RWJ-445380 Administered to Patients With Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alza Corporation, DE, USA (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR012367
Record Dates: First submitted 2006-11-03; First posted 2006-11-07 (Estimated); Last update posted 2011-02-18 (Estimated); Status verified 2011-02

CONDITIONS: Chronic Small Plaque Psoriasis
Keywords: psoriasis; skin; auto immune
MeSH Terms: conditions — Psoriasis

INTERVENTIONS:
Drug: RWJ-445380

SUMMARY:
The primary objective of the study is to evaluate the safety and tolerability of 50, 100, 200, and 300 mg/day doses of RWJ-445380 for up to 12 weeks in patients with plaque psoriasis

DETAILED DESCRIPTION:
Trials with a new, first-in-class drug will be done to ascertain safety, tolerability, absorption and other effects in the treatment of psoriasis, such as effects on biomarkers. Approximately 60 adult patients with psoriasis covering at least 3 percent of their body surface area will be recruited for the study. They will be randomly assigned to one of 5 treatment arms each patient has an equal chance of receiving the placebo, 50 mg, 100 mg, 200 mg, or 300 mg dose. Patients will receive study medication in a blinded fashion, i.e, the patient, the doctor and the study sponsor will not know what group the patient is in until all patients complete the study. Patients will take the medication daily for 12 weeks. The study will be enrolled in two enrollment groups of about 30 patients each, so that extent of side effects can be ascertained and expectations on their extent confirmed. The investigator and the sponsor will monitor the study for the occurrence of possible side effects. In addition to a screening visit, patients will have visits every week for the first month, and then every two weeks until 12 weeks of treatment. At 12 weeks, there are 2 visits on consecutive days for tests and there is one followup visit 4 weeks after the last dose of study drug is taken.

Medical history, physical examination, blood pressure and heart rate, and ECGs are checked periodically. Blood samples will be taken for standard laboratory tests as well as special tests of the drug blood level, biomarkers to see whether the drug might be affecting the biological pathway of antigen presentation, and skin biopsies from areas both involved and not involved with psoriasis. The blood and skin samples will be used to see whether some of the characteristics of psoriasis are changed by taking the drug. Samples will also be taken to see whether certain types of immune cells are affected by taking the drug. Immunizations with tetanus and hepatitis A vaccines will be done to see if taking the drug might affect immune responses to these agents. Patients will receive RWJ-445380, 50, 100, 200, 300 mg, or placebo. Patients will receive an oral capsule daily for up to 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of plaque psoriasis for at least 6 months
* willingness to undergo tissue biopsies

Exclusion Criteria:

* No current oral or injectable medications for psoriasis (30 days to 3 months)
* no other major health issues

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-09; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of RWJ-445380 for up to 12 weeks; assessing adverse events, vital signs, laboratory assessments, physical exam and ECGs in patients with psoriasis

SECONDARY OUTCOMES:
Explore effectiveness of drug through accepted psoriasis clinical measures and biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Alza Corporation Clinical Trial, Study Director — ALZA